CLINICAL TRIAL: NCT00479934
Title: Phase II Randomized Double Blind Clinical Trial of'Imatinib Mesylate STI571 (Glivec®) Versus Placebo in Patients With Severe Cutaneous Scleroderma or Systemic Sclerosis With Severe Cutaneous Involvement.
Brief Title: Efficacy and Safety of Imatinib in Scleroderma
Acronym: SCLEROGLIVEC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry of Health, France (Other Government); Novartis (Industry)
Responsible Party: Jean-Pierre LEROY / Clinical Research and Innovation Director, University Hospital, Bordeaux
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHUBX 2006/05; 2006/017
Record Dates: First submitted 2007-05-29; First posted 2007-05-30 (Estimated); Last update posted 2011-03-04 (Estimated); Status verified 2011-03

CONDITIONS: Scleroderma, Localized; Scleroderma, Systemic
Keywords: scleroderma; imatinib; PDGFR; Rodnan
MeSH Terms: conditions — Scleroderma, Localized; Scleroderma, Systemic; Scleroderma, Diffuse | interventions — Imatinib Mesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 6 month treatment with Imtinib 400mg/day
  Interventions: Drug: imatinib mesylate
- 2 (Placebo Comparator): 6 month treatment with Placebo 400mg/day
  Interventions: Drug: imatinib mesylate

INTERVENTIONS:
Drug: imatinib mesylate — 6 month treatment with 400mg/day (per os)

SUMMARY:
In vitro studies have shown that imatinib 1mM inhibits strongly the growth of cutaneous fibroblasts. The hypothesis is that imatinib inhibits PDGFR which is known to be a potential target for the molecule, as recently also proposed after the discovery of autoantibodies activating the PDGF receptors. Recent data indicate that TGFb is also a potential target of imatinib. Cutaneous scleroderma is characterized by progressive cutaneous fibrosis caused by hyperactive dermal fibroblasts. Since no established treatment for skin sclerosis in scleroderma is currently available. This study will test the safety and efficacy of imatinib in the treatment of patients with scleroderma and severe cutaneous involvement.

DETAILED DESCRIPTION:
This study will test the efficacy and tolerance of patients with a high score of induration (modified Rodnan score > 20/54) Comparison : 34 patients with severe forms of cutaneous involvement will be evaluated in a double blind RCT comparing imatinib 400mg/j and placebo in a 6 month period. Efficacy will be assessed using a cutaneous induration scale and skin biopsy, and quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old
* Documented diagnostic of scleroderma (systemic or cutaneous)
* Severe cutaneous sclerodermia or systemic sclerodermia with m-Rodnan score > 20/51
* Ejection fraction of more than 45 per cent at cardiac ultrasound pre-inclusion study
* Woman with efficient contraceptive method during trail treatment and during 3 month after the end of trial treatment
* All female patients with reproductive potential must have a negative pregnancy test (serum or urine) within the 7 days prior to enrolment
* Affiliated or profit patient of a social security system
* Signed informed consent

Exclusion Criteria:

* new systemic treatment, potentially interfering with disease progression, beginning 3 months prior the start trial treatment
* Patient with isolated cutaneous scleroderma treated with a drug potentially interfering with the course of the disease 4 weeks before starting the trial (Systemic corticosteroids, methotrexate, cyclophosphamide, bosentan)
* Scleroderma " en coup de sabre "
* Severe organ failure or anomaly of blood chemistry/hematology (bilirubin, SGOT, SGPT, creatinine > 1,5 ´ upper normal limit, polymorphonuclear granulocytes less than 1*10*9/l or platelets less than 50*10*9/l),
* Ongoing cancer
* Ejection fraction ≤ 45 per cent at cardiac ultrasound pre inclusion study
* myocardial infarction of less than 6 mois at pre inclusion visit
* Non controlled chronic illness (diabetes, chronic kidney failure, chronic hepatitis, HIV infection),
* Major surgery less than two weeks before inclusion
* Pregnancy or lactation
* Absence of validated contraception in childbearing women.
* Contraindication to imatinib mesylate treatment as specified in product specifications
* Non observance anticipated and absence of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-12; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Compare the efficacy of imatinib mesylate vs placebo based on the percent variation of modified Rodnan score (0-51) between inclusion and 6-month visits. | 6 month

SECONDARY OUTCOMES:
Compare efficacy of imatinib mesylate vs placebo based on the percent variation of modified Rodnan score between the inclusion and the various time points of follow-up. | 1, 3 and 12 month
Assess skin thickness at inclusion and at 6 months using skin biopsies | 6 month
Assessment of quality of life using DLQI (Dermatology Quality of Life Index) and HAQ (Health Assessment Questionnaire). | At 1, 3, 6 month and 1 year,
Assess tolerance of treatment (clinical and laboratory monitoring of side effects) | All along the trial
Assess effects of treatment on non cutaneous symptoms in systemic sclerosis patients | All along the trial

CONTACTS AND LOCATIONS:
Overall Officials: Alain TAIEB, Pr., Study Director — University Hospital, Bordeaux, France; Geneviève CHENE, Pr, Study Chair — University Hospital, Bordeaux, France; Alian TAIEB, Pr., Principal Investigator — University Hospital, Bordeaux, France
Locations (12):
- France (12):
  - Service de Dermatologie et services de médecine interne et vasculaire - Hôpital St André - CHU de Bordeaux, Bordeaux
  - Service de Rhumatologie, Hôpital Pellegrin-Tondu CHU de Bordeaux, Bordeaux
  - Service de Dermatologie - CHG Libourne, Libourne
  - Service de dermatologie - CHU de Limoges, Limoges
  - Service de Médecin interne - Hôpital central, Nancy
  - Service de Médecine interne - Hôpital Saint Louis, Paris
  - Service de Dermatologie - service de médecine interne et vasculaire - hopital haut Lévêque - av.de magellan, Pessac
  - Service de Dermatologie - CHG Périgueux, Périgueux
  - Service de Rhumatologie - CHU de Strasbourg, Strasbourg
  - Service de Dermatologie - CHU de Toulouse - Hopital Purpan, Toulouse
  - Service de Médecine interne - CHU de Tours, Tours
  - Néphrologie et Médecine interne - CH de Valenciennes, Valenciennes